CLINICAL TRIAL: NCT00638794
Title: Assessment of Dual AntiPlatelet Therapy With Drug Eluting Stents
Acronym: ADAPT-DES
Status: Completed | Type: Observational
Sponsor: Cardiovascular Research Foundation, New York (Other)
Collaborators: Dickson Advanced Analytics Group (Unknown)
Responsible Party: Sponsor
Other Study IDs: ADAPT-DES
Record Dates: First submitted 2008-02-28; First posted 2008-03-19 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2012-08

CONDITIONS: Coronary Artery Disease
Keywords: Myocardial Infarction; Myocardial Ischemia
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction; Myocardial Ischemia | interventions — Drug-Eluting Stents

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Surgical: Patients with coronary artery disease undergoing stent-assisted percutaneous coronary intervention (PCI) using DES without major procedural complications.
- Observational: Consecutive patients with coronary artery disease undergoing stent-assisted percutaneous coronary intervention (PCI) using DES without major procedural complications
  Interventions: Device: Drug -Eluting Stent (Taxus™, Cypher®, Endeavor™, Xience V™)

INTERVENTIONS:
Device: Drug -Eluting Stent (Taxus™, Cypher®, Endeavor™, Xience V™) — PCI using any FDA approved drug-eluting stent; Taxus Express2 - Paclitaxel-Eluting Coronary Stent System Cypher Sirolimus-eluting coronary stent Endeavor ABT-578 Eluting Coronary Stent System Xience V Everolimus Eluting Coronary Stent System
  Other Names: Taxus™, Cypher®, Endeavor™, Xience V™
  Groups: Observational

SUMMARY:
Prospective, multicenter, registry of at least 11,000 (and up to 15,000) consecutive patients with coronary artery disease undergoing stent-assisted percutaneous coronary intervention (PCI) using DES without major procedural complications.

DETAILED DESCRIPTION:
To determine:

1. the frequency, timing and correlates (clinical and angiographic) of drug-eluting stent (DES) thrombosis in a patient population with few clinical and angiographic exclusion criteria,
2. the relationship of aspirin and/or clopidogrel hyporesponsiveness, and general platelet reactivity to early and late DES thrombosis in separate phases stratified by whether the patient is taking dual (aspirin plus clopidogrel) or single (aspirin alone) antiplatelet therapy, and
3. combining the findings from the above 2 objectives, to identify a cohort representing a significant proportion of all patients at increased risk to have early and/or late DES stent thrombosis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing PCI in whom at least one DES is implanted and in whom PCI of all treated lesions is successful (diameter stenosis <30% with TIMI 3 flow in all treated lesions) without major complications (defined as freedom from procedural death, intra-procedural stent thrombosis, procedural myocardial infarction or sustained vessel closure, or need for emergency bypass graft surgery). One or more bare metal stents (BMS) may be implanted, and other lesions may be treated without stenting as long as at least one DES is implanted. However, the procedure must be successful and uncomplicated (as defined above) for all lesions (DES + BMS + non-stent).
2. Aspirin use: Adequate aspirin loading given prior to PCI: at least 300 mg non enteric coated oral aspirin at least 1 hour prior to the procedure or 324 mg chewed or 250 mg IV aspirin at least 30 minutes prior to the procedure.
3. Patient has Hematocrit between 30 and 52% and Platelet Count greater than 100,000/µl.
4. For US sites: Only FDA-approved DES stents may be used in this study. For OUS sites: Only DES stents that are CE marked for approval may be used in this study.
5. PCI performed with unfractionated or low molecular weight heparin, or bivalirudin as the procedural antithrombin.
6. Patient or guardian able to provide informed written consent.

Exclusion Criteria:

1. Patients in whom blood for Accumetrics VerifyNow platelet function testing cannot be drawn after the minimum clopidogrel loading duration and Glycoprotein (GP) IIb/IIIa inhibitor washout duration as follows:

   1. Clopidogrel loading: Clopidogrel loading pre PCI is recommended, but post PCI clopidogrel loading is acceptable per standard of care. In all patients (whether or not clopidogrel is initiated pre or post PCI), prior to blood drawing for VerifyNow platelet function testing, a 600 mg loading dose must have been given at least 6 hours prior, or a 300 mg loading dose must have been given at least 12 hours prior, or the patient must have been maintained on at least 75 mg of clopidogrel daily for at least 5 days.
   2. GP IIb/IIIa inhibitor washout: Eptifibatide or tirofiban must have been discontinued for at least 24 hours prior to VerifyNow platelet function testing. Abciximab must have been discontinued for at 10 days prior to VerifyNow platelet function testing.
2. Inability of the VerifyNow system to measure either Aspirin, P2Y12 or IIb/IIIa platelet responsiveness.
3. Severe allergy to stainless steel, contrast dye, all anti-thrombin agents (unfractionated and low molecular weight heparin and bivalirudin), aspirin or clopidogrel that cannot be adequately pre-medicated.
4. Concurrent enrollment in another trial that involves an investigational stent, antithrombotic or antiplatelet agent. Patient in other investigational trials that have not reached their primary endpoint may be enrolled in ADAPT-DES as long as the other trials do not involve an investigational stent, antithrombotic or antiplatelet agent and inclusion of such patient will have no effect on the endpoint of either study.
5. Patients in whom bypass graft surgery is planned within 2 years.
6. Patients with stent thrombosis before the performance of pre-discharge VerifyNow platelet function testing.
7. Patients unwilling or unable to complete clinical follow-up for the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient undergoing PCI in whom at least one DES is implanted and in whom PCI of all treated lesions is successful (diameter stenosis <30% with TIMI 3 flow in all treated lesions) without major complications (defined as freedom from procedural death, intraprocedural stent thrombosis, procedural myocardial infarction or sustained vessel closure, or need for emergency bypass graft surgery).
Sampling Method: Probability Sample
Enrollment: 8575 (Actual)
Dates: Start 2008-01; Primary Completion 2011-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Definite or probable stent thrombosis using the Academic Research Consortium (ARC) definition, primary events only. | 30 days, 1 year, 2 year

SECONDARY OUTCOMES:
ARC definite, probable, possible or any stent thrombosis, utilizing primary only and then primary + secondary thromboses; death, MI, recurrent ischemia necessitating repeat target lesion and target vessel intervention and MACE. | 1 day, 30 days, 1 year, 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Gregg W. Stone, MD, Principal Investigator — CardioVascular Research Foundation
Locations (8):
- United States (8):
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Columbia University Medical Center & New York Presbyterian, New York, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - LeBauer Cardiovascular Research, Greensboro, North Carolina
  - FirstHealth Moore Regional Hospital, Pinehurst, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - Lehigh Valley Hospital and Health Network, Allentown, Pennsylvania
  - Wellmont Holston Valley Medical Center, Kingsport, Tennessee

REFERENCES:
- [Derived] Shahim B, Redfors B, Stuckey TD, Liu M, Zhou Z, Witzenbichler B, Weisz G, Rinaldi MJ, Neumann FJ, Metzger DC, Henry TD, Cox DA, Duffy PL, Brodie BR, Srdanovic I, Madhavan MV, Mazzaferri EL Jr, Mehran R, Ben-Yehuda O, Kirtane AJ, Stone GW. On-Treatment Platelet Reactivity and Ischemic Outcomes in Patients With Diabetes Mellitus: Two-Year Results From ADAPT-DES. J Am Heart Assoc. 2023 Jan 3;12(1):e026482. doi: 10.1161/JAHA.122.026482. Epub 2022 Dec 24. PMID 36565189
- [Derived] Redfors B, Kirtane AJ, Liu M, Musikantow DR, Witzenbichler B, Rinaldi MJ, Metzger DC, Weisz G, Stuckey TD, Brodie BR, Ben-Yehuda O, Mehran R, Stone GW. Dual Antiplatelet Therapy Discontinuation, Platelet Reactivity, and Adverse Outcomes After Successful Percutaneous Coronary Intervention. JACC Cardiovasc Interv. 2022 Apr 25;15(8):797-806. doi: 10.1016/j.jcin.2022.01.300. PMID 35450679
- [Derived] Gupta R, Kirtane AJ, Liu Y, Crowley A, Witzenbichler B, Rinaldi MJ, Metzger DC, Weisz G, Stuckey TD, Brodie BR, Mehran R, Ben-Yehuda O, Stone GW. Impact of Smoking on Platelet Reactivity and Clinical Outcomes After Percutaneous Coronary Intervention: Findings From the ADAPT-DES Study. Circ Cardiovasc Interv. 2019 Nov;12(11):e007982. doi: 10.1161/CIRCINTERVENTIONS.119.007982. Epub 2019 Nov 1. PMID 31672031
- [Derived] Maehara A, Mintz GS, Witzenbichler B, Weisz G, Neumann FJ, Rinaldi MJ, Metzger DC, Henry TD, Cox DA, Duffy PL, Brodie BR, Stuckey TD, Mazzaferri EL Jr, McAndrew T, Genereux P, Mehran R, Kirtane AJ, Stone GW. Relationship Between Intravascular Ultrasound Guidance and Clinical Outcomes After Drug-Eluting Stents. Circ Cardiovasc Interv. 2018 Nov;11(11):e006243. doi: 10.1161/CIRCINTERVENTIONS.117.006243. PMID 30571206
- [Derived] Giustino G, Redfors B, Kirtane AJ, Mehran R, Dangas GD, Witzenbichler B, Neumann FJ, Weisz G, Genereux P, Maehara A, McAndrew T, Farhan S, Rinaldi MJ, Metzger DC, Henry TD, Cox DA, Duffy PL, Mazzaferri EL Jr, Brodie BR, Stuckey TD, Gurbel P, Ben-Yehuda O, Stone GW. Platelet Reactivity and Risk of Ischemic Stroke After Coronary Drug-Eluting Stent Implantation: From the ADAPT-DES Study. JACC Cardiovasc Interv. 2018 Jul 9;11(13):1277-1286. doi: 10.1016/j.jcin.2018.01.263. Epub 2018 Jun 13. PMID 29908967
- [Derived] Redfors B, Genereux P, Witzenbichler B, Kirtane AJ, McAndrew T, Weisz G, Stuckey TD, Henry TD, Maehara A, Mehran R, Stone GW. Bleeding Severity After Percutaneous Coronary Intervention. Circ Cardiovasc Interv. 2018 Mar;11(3):e005542. doi: 10.1161/CIRCINTERVENTIONS.117.005542. PMID 29870382
- [Derived] Redfors B, Genereux P, Witzenbichler B, McAndrew T, Diamond J, Huang X, Maehara A, Weisz G, Mehran R, Kirtane AJ, Stone GW. Percutaneous Coronary Intervention of Saphenous Vein Graft. Circ Cardiovasc Interv. 2017 May;10(5):e004953. doi: 10.1161/CIRCINTERVENTIONS.117.004953. PMID 28495896
- [Derived] Gupta R, Kirtane AJ, Ozan MO, Witzenbichler B, Rinaldi MJ, Metzger DC, Weisz G, Stuckey TD, Brodie BR, Mehran R, Ben-Yehuda O, Stone GW. Platelet Reactivity and Clinical Outcomes After Coronary Artery Implantation of Drug-Eluting Stents in Subjects With Peripheral Arterial Disease: Analysis From the ADAPT-DES Study (Assessment of Dual Antiplatelet Therapy With Drug-Eluting Stents). Circ Cardiovasc Interv. 2017 Mar;10(3):e004904. doi: 10.1161/CIRCINTERVENTIONS.116.004904. PMID 28288963
- [Derived] Yu J, Mehran R, Baber U, Ooi SY, Witzenbichler B, Weisz G, Rinaldi MJ, Neumann FJ, Metzger DC, Henry TD, Cox DA, Duffy PL, Mazzaferri EL Jr, Brodie BR, Stuckey TD, Maehara A, Xu K, Ben-Yehuda O, Kirtane AJ, Stone GW. Sex Differences in the Clinical Impact of High Platelet Reactivity After Percutaneous Coronary Intervention With Drug-Eluting Stents: Results From the ADAPT-DES Study (Assessment of Dual Antiplatelet Therapy With Drug-Eluting Stents). Circ Cardiovasc Interv. 2017 Feb;10(2):e003577. doi: 10.1161/CIRCINTERVENTIONS.116.003577. PMID 28193677
- [Derived] Wang B, Mintz GS, Witzenbichler B, Souza CF, Metzger DC, Rinaldi MJ, Duffy PL, Weisz G, Stuckey TD, Brodie BR, Matsumura M, Yamamoto MH, Parvataneni R, Kirtane AJ, Stone GW, Maehara A. Predictors and Long-Term Clinical Impact of Acute Stent Malapposition: An Assessment of Dual Antiplatelet Therapy With Drug-Eluting Stents (ADAPT-DES) Intravascular Ultrasound Substudy. J Am Heart Assoc. 2016 Dec 22;5(12):e004438. doi: 10.1161/JAHA.116.004438. PMID 28007741
- [Derived] Kobayashi N, Mintz GS, Witzenbichler B, Metzger DC, Rinaldi MJ, Duffy PL, Weisz G, Stuckey TD, Brodie BR, Parvataneni R, Kirtane AJ, Stone GW, Maehara A. Prevalence, Features, and Prognostic Importance of Edge Dissection After Drug-Eluting Stent Implantation: An ADAPT-DES Intravascular Ultrasound Substudy. Circ Cardiovasc Interv. 2016 Jul;9(7):e003553. doi: 10.1161/CIRCINTERVENTIONS.115.003553. PMID 27402854
- [Derived] Yun KH, Mintz GS, Witzenbichler B, Inaba S, Shimizu T, Metzger DC, Rinaldi MJ, Mazzaferri EL Jr, Duffy PL, Weisz G, Stuckey TD, Brodie BR, Kirtane AJ, Stone GW, Maehara A. Relationship Between Platelet Reactivity and Culprit Lesion Morphology: An Assessment From the ADAPT-DES Intravascular Ultrasound Substudy. JACC Cardiovasc Imaging. 2016 Jul;9(7):849-854. doi: 10.1016/j.jcmg.2015.08.019. Epub 2016 Feb 17. PMID 26897675
- [Derived] Kirtane AJ, Parikh PB, Stuckey TD, Xu K, Witzenbichler B, Weisz G, Rinaldi MJ, Neumann FJ, Metzger DC, Henry TD, Cox DA, Duffy PL, Brodie BR, Mazzaferri EL Jr, Parvataneni R, Maehara A, Genereux P, Mehran R, Stone GW. Is There an Ideal Level of Platelet P2Y12-Receptor Inhibition in Patients Undergoing Percutaneous Coronary Intervention?: "Window" Analysis From the ADAPT-DES Study (Assessment of Dual AntiPlatelet Therapy With Drug-Eluting Stents). JACC Cardiovasc Interv. 2015 Dec 28;8(15):1978-1987. doi: 10.1016/j.jcin.2015.08.032. PMID 26738669
- [Derived] Dohi T, Maehara A, Witzenbichler B, Rinaldi MJ, Mazzaferri EL Jr, Duffy PL, Weisz G, Neumann FJ, Henry TD, Cox DA, Stuckey TD, Brodie BR, Litherland C, Brener SJ, Kirtane AJ, Mintz GS, Stone GW. Etiology, Frequency, and Clinical Outcomes of Myocardial Infarction After Successful Drug-Eluting Stent Implantation: Two-Year Follow-Up From the ADAPT-DES Study. Circ Cardiovasc Interv. 2015 Dec;8(12):e002447. doi: 10.1161/CIRCINTERVENTIONS.114.002447. PMID 26643737
- [Derived] Brodie BR, Garg A, Stuckey TD, Kirtane AJ, Witzenbichler B, Maehara A, Weisz G, Rinaldi MJ, Neumann FJ, Metzger DC, Mehran R, Parvataneni R, Stone GW. Fixed and Modifiable Correlates of Drug-Eluting Stent Thrombosis From a Large All-Comers Registry: Insights From ADAPT-DES. Circ Cardiovasc Interv. 2015 Oct;8(10):e002568. doi: 10.1161/CIRCINTERVENTIONS.114.002568. PMID 26415600
- [Derived] Genereux P, Giustino G, Witzenbichler B, Weisz G, Stuckey TD, Rinaldi MJ, Neumann FJ, Metzger DC, Henry TD, Cox DA, Duffy PL, Mazzaferri E, Yadav M, Francese DP, Palmerini T, Kirtane AJ, Litherland C, Mehran R, Stone GW. Incidence, Predictors, and Impact of Post-Discharge Bleeding After Percutaneous Coronary Intervention. J Am Coll Cardiol. 2015 Sep 1;66(9):1036-45. doi: 10.1016/j.jacc.2015.06.1323. PMID 26314532
- [Derived] Petersen JE, Bouwens EA, Tamayo I, Turner L, Wang CW, Stins M, Theander TG, Hermida J, Mosnier LO, Lavstsen T. Protein C system defects inflicted by the malaria parasite protein PfEMP1 can be overcome by a soluble EPCR variant. Thromb Haemost. 2015 Nov;114(5):1038-48. doi: 10.1160/TH15-01-0018. Epub 2015 Jul 9. PMID 26155776
- [Derived] Baber U, Mehran R, Kirtane AJ, Gurbel PA, Christodoulidis G, Maehara A, Witzenbichler B, Weisz G, Rinaldi MJ, Metzger DC, Henry TD, Cox DA, Duffy PL, Mazzaferri EL Jr, Xu K, Parise H, Brodie BR, Stuckey TD, Stone GW. Prevalence and impact of high platelet reactivity in chronic kidney disease: results from the Assessment of Dual Antiplatelet Therapy with Drug-Eluting Stents registry. Circ Cardiovasc Interv. 2015 Jun;8(6):e001683. doi: 10.1161/CIRCINTERVENTIONS.115.001683. PMID 26056248
- [Derived] Kang SJ, Mintz GS, Witzenbichler B, Metzger DC, Rinaldi MJ, Duffy PL, Weisz G, Stuckey TD, Brodie BR, Shimizu T, Xu K, Kirtane AJ, Stone GW, Maehara A. Effect of obesity on coronary atherosclerosis and outcomes of percutaneous coronary intervention: grayscale and virtual histology intravascular ultrasound substudy of assessment of dual antiplatelet therapy with drug-eluting stents. Circ Cardiovasc Interv. 2014 Dec 31;8(1):e001392. doi: 10.1161/CIRCINTERVENTIONS.114.001392. Print 2015 Jan. PMID 25552564
- [Derived] Witzenbichler B, Maehara A, Weisz G, Neumann FJ, Rinaldi MJ, Metzger DC, Henry TD, Cox DA, Duffy PL, Brodie BR, Stuckey TD, Mazzaferri EL Jr, Xu K, Parise H, Mehran R, Mintz GS, Stone GW. Relationship between intravascular ultrasound guidance and clinical outcomes after drug-eluting stents: the assessment of dual antiplatelet therapy with drug-eluting stents (ADAPT-DES) study. Circulation. 2014 Jan 28;129(4):463-70. doi: 10.1161/CIRCULATIONAHA.113.003942. Epub 2013 Nov 26. PMID 24281330
- [Derived] Stone GW, Witzenbichler B, Weisz G, Rinaldi MJ, Neumann FJ, Metzger DC, Henry TD, Cox DA, Duffy PL, Mazzaferri E, Gurbel PA, Xu K, Parise H, Kirtane AJ, Brodie BR, Mehran R, Stuckey TD; ADAPT-DES Investigators. Platelet reactivity and clinical outcomes after coronary artery implantation of drug-eluting stents (ADAPT-DES): a prospective multicentre registry study. Lancet. 2013 Aug 17;382(9892):614-23. doi: 10.1016/S0140-6736(13)61170-8. Epub 2013 Jul 26. PMID 23890998